CLINICAL TRIAL: NCT05968937
Title: Baclofen in Chronic Pelvic Pain, a Randomized, Double-Blind, Placebo Controlled Trial
Brief Title: Vaginal Baclofen Suppositories in Chronic Pelvic Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Ankita Gupta, Principal Investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22.1000
Record Dates: First submitted 2023-05-12; First posted 2023-08-01 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: Baclofen; vaginal suppository; pelvic floor muscle dysfunction

STUDY DESIGN:
Intervention Model Description: This is a single-center, double-blinded, placebo-controlled, randomized trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be carried out by a computer-based algorithm that will generate study/subject number. This number will correspond with treatment and communicate to The Louisville compounding pharmacy the appropriate drug to distribute without the unblinding of patient or provider. with a stratified block randomization scheme (with a random block size of 4, 6, and 8 participants). Randomization will be stratified based on pelvic muscle tenderness on exam - stratifying by 0-5/10 and 6-10/10 tenderness of pelvic floor musculature on physical exam
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vaginal baclofen suppository (Active Comparator): Baclofen 20mg in Supposibase F vaginal suppository daily per vagina
  Interventions: Drug: 20 mg baclofen vaginal suppository daily per vagina
- Vaginal placebo suppository (Placebo Comparator): Supposibase F vaginal suppository daily per vagina
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 20 mg baclofen vaginal suppository daily per vagina — 20 mg baclofen vaginal suppository in Supposibase F daily per vagina - to be compounded by The Louisville Compounding Pharmacy
  Arms: Vaginal baclofen suppository
Drug: Placebo — Vaginal suppository composed of Supposibase F daily per vagina
  Arms: Vaginal placebo suppository

SUMMARY:
The purpose of this study is to evaluate if baclofen vaginal suppositories improve symptoms of Chronic Pelvic Pain (CPP).

Participants in this study will take four short questionnaires prior to being randomized. Randomization is like flipping a coin; participants have an equal likelihood of being randomized to the treatment group (vaginal baclofen suppositories) or placebo group (vaginal suppository without baclofen ingredient). Participants will take their assigned treatment nightly for 8 weeks. Follow up visits will be at the 4 and 8 week time frames, when questionnaires will again be completed. Participants may receive additional treatments for CPP during the course of the study. After 8 weeks Participants will be offered a prescription for baclofen suppositories and the study drug will be stopped. Follow up on patient symptoms with questionnaires will again occur at 12 weeks.

DETAILED DESCRIPTION:
Study Design/Methodology

This is a single center, double-blinded, placebo-controlled, randomized trial. Women will be recruited from a subspecialty clinic at the University of Louisville and be eligible for participation if they meet the diagnosis of Chronic Pelvic Pain and are between the ages of 18-65 years old. Eligible, consenting participants will undergo randomization with equal probability of assignment to one of the two groups:

1. Baclofen 20mg vaginal suppository daily per vagina and
2. placebo.

Participants will be blinded to study allocation. Baclofen or placebo suppositories will be continued to 8 weeks, at which time all participants will be offered a baclofen suppository prescription. Patients will then follow up at the 12 week mark and whether they continued baclofen suppositories and pill count will be recorded in addition to the below questionnaires.

Clinical outcomes and questionnaires will be assessed at baseline and after 4, 8, and 12 weeks of treatment. Participants will be randomized with a stratified block randomization scheme (with a random block size of 4, 6, and 8 participants).

Participants will be required to come in for at least 1 visit at 8 weeks to assess pelvic muscle dysfunction and perform pill count.

We hypothesize a significant change in PROMIS Pain Interference score, patient satisfaction, PROMIS global health scores, and PROMIS sexual function scores for patients assigned to the baclofen treatment arm.

Inclusion Criteria:

* Women ages 18-65 years old
* Women are not sexually active, sexually active with same sex partners or are on effective contraception
* Diagnosed with Chronic Pelvic Pain

Exclusion Criteria:

* Gross hematuria
* Currently pregnant or breastfeeding
* Unable to speak and read English
* History of allergic reaction to baclofen tablet
* History of allergic reaction to components of placebo (coconut oil)
* History of gastrointestinal, genitourinary, or pelvic cancer in the last 5 years

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-65 years old
* Women are not sexually active, sexually active with same sex partners or are on effective contraception
* Diagnosed with Chronic Pelvic Pain

Exclusion Criteria:

* Gross hematuria
* Currently pregnant or breastfeeding
* Unable to speak and read English
* History of allergic reaction to baclofen tablet
* History of allergic reaction to components of placebo (coconut oil)
* History of gastrointestinal, genitourinary, or pelvic cancer in the last 5 years

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogue Score (VAS) 1-100 for pain | at 8 weeks of suppository use
  VAS is a 1-100mm scale with lower scores indicating less pain

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference score | at baseline and at 4, 8 and 12 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) pain interference score is a 40-200 point scale with lower values indicating lower pain interference with quality of life
Pelvic floor impact questionnaire | at baseline and at 4, 8, and 12 week follow up
  pelvic floor impact questionnaire is a 0-63 point composite scale consisting of questions concerning bladder/urinary, bowel/rectal, and vaginal/pelvic symptoms with higher values indicating higher symptoms
Pelvic floor disability index (PFDI) questionnaire | at baseline and at 4, 8, and 12 week follow up
  the pelvic floor disability index (PFDI) questionnaire is a composite questionnaire on a 0-80 point scale containing questions regarding pelvic organ prolapse, colorectal/anal distress, and urinary distress questions with higher scores indicating higher symptoms
Visual analogue Score (VAS) 1-100 for pain | at baseline and at 4 and 12 week follow up
  VAS is a 1-100mm scale with lower scores indicating less pain
O'Leary Sant questionnaire | at baseline and at 4, 8, and 12 week follow up
  O'Leary Sant questionnaire is a 0 to 37 point score with higher points indicating increased symptoms
Patient-Reported Outcomes Measurement Information System (PROMIS) global health score | at baseline and at 4, 8, and 12 week follow up
  Patient-Reported Outcomes Measurement Information System (PROMIS) global health score is a 9-45 point scale with higher scores indicating better overall health and quality of life
Overall Satisfaction | at 4, 8, and 12 week follow up
  Overall Satisfaction is a yes/no questionnaire with if "yes" is selected one selects choices from "somewhat" to "quite a bit" in satisfaction. "quite a bit" would indicate greater satisfaction.
Patient-Reported Outcomes Measurement Information System (PROMIS) Sexual function score | at 0, 4, 8, and 12 week follow up
  Patient-Reported Outcomes Measurement Information System (PROMIS) Sexual function score is a 9-36 point score with higher scores indicating higher bother related to sexual function
Number of other treatments for chronic pelvic pain during the trial period | at 4, 8, and 12 week follow up
  Number of other treatments for chronic pelvic pain during the trial period to determine if results are clouded by other, appropriate, evidence based treatments received for chronic pelvic pain.
Pill Count | at 4, 8, and 12 week follow up
  Pill Count to determine how many doses of the study medication have been missed

CONTACTS AND LOCATIONS:
Overall Officials: Rodger W Rothenberger, MD, Study Director — University of Louisville
Locations (1):
- ULP Female Pelvic Medicine and Reconstructive Surgery - Springs Medical Center Suite 190, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
This study information will be sourced from the subjects. Identifying information and data collected during this study will be kept secure and confidential. For confidentiality, only research team members will have access to the study information in the database. Subjects will be assigned a unique study ID that will be used on all case report forms and database reporting. The database that will be used is REDCap which is HIPPA (Health Insurance Portability and Accountability Act of 1996) compliant, encrypted, and password protected. Any hard copies will be maintained in a locked cabinet in a locked office by a member of the research team.
  The research personnel in this study are CITI and HIPAA trained. If new research personnel are added, an amendment will be submitted to and approved by the IRB before being allowed to participate in the study

REFERENCES:
- [Background] Doggweiler R, Whitmore KE, Meijlink JM, Drake MJ, Frawley H, Nordling J, Hanno P, Fraser MO, Homma Y, Garrido G, Gomes MJ, Elneil S, van de Merwe JP, Lin ATL, Tomoe H. A standard for terminology in chronic pelvic pain syndromes: A report from the chronic pelvic pain working group of the international continence society. Neurourol Urodyn. 2017 Apr;36(4):984-1008. doi: 10.1002/nau.23072. Epub 2016 Aug 26. PMID 27564065
- [Background] Lamvu G, Carrillo J, Ouyang C, Rapkin A. Chronic Pelvic Pain in Women: A Review. JAMA. 2021 Jun 15;325(23):2381-2391. doi: 10.1001/jama.2021.2631. PMID 34128995
- [Background] Chronic Pelvic Pain: ACOG Practice Bulletin, Number 218. Obstet Gynecol. 2020 Mar;135(3):e98-e109. doi: 10.1097/AOG.0000000000003716. PMID 32080051
- [Background] Mathias SD, Kuppermann M, Liberman RF, Lipschutz RC, Steege JF. Chronic pelvic pain: prevalence, health-related quality of life, and economic correlates. Obstet Gynecol. 1996 Mar;87(3):321-7. doi: 10.1016/0029-7844(95)00458-0. PMID 8598948
- [Background] Brawn J, Morotti M, Zondervan KT, Becker CM, Vincent K. Central changes associated with chronic pelvic pain and endometriosis. Hum Reprod Update. 2014 Sep-Oct;20(5):737-47. doi: 10.1093/humupd/dmu025. Epub 2014 Jun 11. PMID 24920437
- [Background] Shafrir AL, Martel E, Missmer SA, Clauw DJ, Harte SE, As-Sanie S, Sieberg CB. Pelvic floor, abdominal and uterine tenderness in relation to pressure pain sensitivity among women with endometriosis and chronic pelvic pain. Eur J Obstet Gynecol Reprod Biol. 2021 Sep;264:247-253. doi: 10.1016/j.ejogrb.2021.07.029. Epub 2021 Jul 22. PMID 34340095
- [Background] Messelink B, Benson T, Berghmans B, Bo K, Corcos J, Fowler C, Laycock J, Lim PH, van Lunsen R, a Nijeholt GL, Pemberton J, Wang A, Watier A, Van Kerrebroeck P. Standardization of terminology of pelvic floor muscle function and dysfunction: report from the pelvic floor clinical assessment group of the International Continence Society. Neurourol Urodyn. 2005;24(4):374-80. doi: 10.1002/nau.20144. No abstract available. PMID 15977259
- [Background] Moldwin RM, Fariello JY. Myofascial trigger points of the pelvic floor: associations with urological pain syndromes and treatment strategies including injection therapy. Curr Urol Rep. 2013 Oct;14(5):409-17. doi: 10.1007/s11934-013-0360-7. PMID 23943509
- [Background] Frederice CP, Brito LGO, Pereira GMV, Lunardi ALB, Juliato CRT. Interventional treatment for myofascial pelvic floor pain in women: systematic review with meta-analysis. Int Urogynecol J. 2021 May;32(5):1087-1096. doi: 10.1007/s00192-021-04725-x. Epub 2021 Feb 27. PMID 33640993
- [Background] Stone RH, Abousaud M, Abousaud A, Kobak W. A Systematic Review of Intravaginal Diazepam for the Treatment of Pelvic Floor Hypertonic Disorder. J Clin Pharmacol. 2020 Dec;60 Suppl 2:S110-S120. doi: 10.1002/jcph.1775. PMID 33274514
- [Background] Juergens S. Alprazolam and diazepam: addiction potential. J Subst Abuse Treat. 1991;8(1-2):43-51. doi: 10.1016/0740-5472(91)90026-7. PMID 2051498
- [Background] Das S, Palappalllil DS, Purushothaman ST, Rajan V. An Unusual Case of Baclofen Abuse. Indian J Psychol Med. 2016 Sep-Oct;38(5):475-476. doi: 10.4103/0253-7176.191383. PMID 27833235
- [Background] Meister MR, Sutcliffe S, Ghetti C, Chu CM, Spitznagle T, Warren DK, Lowder JL. Development of a standardized, reproducible screening examination for assessment of pelvic floor myofascial pain. Am J Obstet Gynecol. 2019 Mar;220(3):255.e1-255.e9. doi: 10.1016/j.ajog.2018.11.1106. Epub 2018 Dec 7. PMID 30527941
- [Background] Amtmann D, Kim J, Chung H, Askew RL, Park R, Cook KF. Minimally important differences for Patient Reported Outcomes Measurement Information System pain interference for individuals with back pain. J Pain Res. 2016 Apr 27;9:251-5. doi: 10.2147/JPR.S93391. eCollection 2016. PMID 27175093